CLINICAL TRIAL: NCT06934902
Title: Attentional Capture by Real-life Episodic Information
Acronym: EPICAPTURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL25_0108
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Healthy Volunteers; Attentional Capture
Keywords: Healthy volunteers; Attentional capture; real-life episodic information

STUDY DESIGN:
Intervention Model Description: Our main hypothesis concerning the role of personal past experiences in guiding spatial attention via the dorsal and ventral attention control system (DAN/VAN) will be tested in two fMRI studies in healthy participants. The use of mobile-mobile technology will allow us to control the formation of episodic memory traces in the real-world. In the testing phase, eye-tracking will permit us to assess the allocation of spatial attention, and fMRI will assess the activation of the attention systems as a function of condition (gaze/attention towards elements associated with previous personal experiences, i.e. pictures of old/seen objects or places, vs. pictures of new/unseen objects/places).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Old vs new objects (Experimental): The following week after the "Old vs new objects" encoding phase of 3 weeks, participants will have an fMRI.
  During fMRI, participants will see objects already seen or not seen during the encoding phase.
  Interventions: Behavioral: Old vs new objects" encoding phase and fMRI
- incongruent vs. congruent contexts (Experimental): The following week after the "incongruent vs. congruent contexts" encoding phase of 3 weeks, participants will have an fMRI.
  During fMRI, participants will see objects encoding in congruent or incongruent contexts.
  Interventions: Behavioral: " incongruent vs. congruent contexts " encoding phase and fMRI

INTERVENTIONS:
Behavioral: Old vs new objects" encoding phase and fMRI — During the encoding phase, a set of 60 objects will be presented to the participants in their everyday life. Pictures of objects sent to their app mobile phone over a period of 3 weeks.
  The following week, participants will have an fMRI. During fMRI, participants will see objects already seen or not seen during the encoding phase.
  Arms: Old vs new objects
Behavioral: " incongruent vs. congruent contexts " encoding phase and fMRI — During the encoding phase, a set of 60 objects will be presented to the participants in their everyday life. Pictures of objects sent to their app mobile phone over a period of 3 weeks. This time, the objects will be chosen according to the participant's location.
  The following week, participants will have an fMRI. During fMRI, participants will see objects encoding in congruent/incongruent contexts.
  Arms: incongruent vs. congruent contexts

SUMMARY:
Attention facilitates the allocation of processing resources and the control of behavior among competing stimuli. Current research focuses primarily on attention control networks in the dorsal frontoparietal (DAN) and ventral (VAN) cortex. However, typical laboratory experiments emphasize task-specific processing, neglecting the possible role of memory. Although a few studies have examined the contribution of memory to attention control, they have generally used simple tasks in the laboratory. These tasks are unlikely to produce true traces of episodic memory, which are - by definition - characterized by complex contextual information (what, where, when) and personal relevance. This research will therefore use an innovative protocol based on mobile phone technology to generate episodes in the participants' real lives and then measure the impact of these past personal experiences on attention allocation (by assessing eye movements) and on the activity of the DAN/VAN system (using functional imaging).

The main hypothesis of the study is that knowledge acquired during everyday life contributes to the subsequent allocation of processing resources, via engagement of the DAN/VAN attention systems.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years old to 40 years old
* Be right-handed
* Do not wear glasses
* Have a mobile-phone compatible with the application, minimum 6rd generation Android operating system, with geo-localization activated and accepted by the user
* Undertake to comply with the instructions and recommendations for MRI examination
* Provide informed written consent to participate in the study

Exclusion Criteria:

* History of known neurological or psychiatric illness
* Cognitive problems limiting the understanding of instructions
* Recent taking psychotropic drugs (antidepressants, anxiolytics, antipsychotics). The main treatments not authorized during this research are the following: Psychotropic treatments (drugs that can induce changes in perception, sensation, mood, consciousness or behavior). Like what:
* Antipsychotics (valproic acid, amisulpride, aripiprazole, clozapine, cyamemazin, haloperidol, loxapine, olanzapine, risperidone).
* Antidepressants (Amitriptyline, Citalopram, Clomipramine, Duloxetine, Escitalopam, Fluoxetine, Mianserine, Mirtazapine, Nortriptyline, Paroxetine, Sertraline, Venlafaxine).
* Anxyolitics
* Pregnant or breastfeeding women
* Persons deprived of their liberty by a judicial or administrative decision
* Persons admitted to a health or social institution for purposes other than research
* Adults subject to a legal protection measure (guardianship, curatorship)
* Persons not affiliated to a social security scheme or beneficiaries of a similar scheme
* Participation in another research study of the current study
* Contraindication for fMRI scanning
* Participant not agreeing to be informed in the event of the incidental discovery of an anomaly on MRI

  • For visit number 2 :
* Alcohol consumption (> 3 drinks) in the 24h before the experiment
* Alcohol consumption the day of the experiment
* Cafeine consumption 1 hour or less before the experiment
* Drug consumption within the 24h preceding the experiment
* Antimalarial treatment within the 3 days preceding the experiment

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
activation pattern in fMRI: "old vs. new" objects (intervention 1) | One time during the week after the 3 weeks encoding phase
  activation pattern in DAN/VAN system in fMRI experiments for the comparison of trials with gaze directed towards "seen/old vs. unseen/new" objects.

SECONDARY OUTCOMES:
activation pattern in fMRI: "place" images in intervention 1 | One time during the week after the 3 weeks encoding phase
  activation pattern in DAN/VAN system in fMRI experiments when participants direct gaze towards the image depicting the location where they were at the time they received an object during the encoding phase, compared with trials when gaze is directed towards the image of a place that was not visited during the encoding phase.
activation pattern in fMRI: incongruent vs. congruent contexts (intervention 2) | One time during the week after the 3 weeks encoding phase
  activation pattern in DAN/VAN system in fMRI experiments for the comparison of trials with gaze directed towards old/seen objects encoded in incongruent vs congruent contexts.

CONTACTS AND LOCATIONS:
Locations (1):
- UCBL1, CRNL Inserm U1028, CNRS UMR5292, équipe IMPACT, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No